CLINICAL TRIAL: NCT03502590
Title: Effectiveness of Airway Control Using the IGEL Laryngeal Mask Airway Device in Patients With Previous Radiotherapy to the Neck
Brief Title: IGEL Laryngeal Mask Airway Device Effectiveness in Irradiated Necks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AC17094
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGEL arm (Experimental): Placement of a physician decided IGEl airway device in patients with prior radiotherapy to the neck to assess adequacy of ventilation
  Interventions: Device: IGEL Laryngeal mask

INTERVENTIONS:
Device: IGEL Laryngeal mask — Insertion of an IGEL device in anaesthetised patients

SUMMARY:
It is known that patients with head and neck cancer who have had radiation therapy to the structures of the neck are at a greater risk of difficult mask ventilation and tracheal intubation than the majority of patients undergoing general anaesthesia.

Failure to maintain oxygenation can lead to catastrophic consequences for any patient undergoing general anaesthesia, such as severe hypoxic brain injury and death.

As such, the current guidelines from the Difficult Airway Society promote the use of a second generation laryngeal mask airway to maintain oxygenation in the event of failed mask ventilation or tracheal intubation, a rescue technique that has in most patient groups a very high chance of success. Unfortunately these guidelines are by necessity generic guidance and do not take into account the clinical performance of these devices in specific patient groups. While there is evidence of the effectiveness of the IGEL device as the primary method of airway maintenance in many studies there are none that describe its clinical performance in a group of patients in whom the rate of failed mask ventilation and tracheal intubation are significantly higher than the general population of patients. It is therefore of great interest to have an idea of the likelihood of success of rescue ventilation with this device in a group of high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Attending for an elective procedure requiring general anaesthesia
* Prior radiotherapy to the neck

Exclusion Criteria:

* General anaesthesia is not the primary airway plan
* Previously known difficult intubation
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Successful insertion of the device and ventilation of the patient | 10 minutes
  Time to successful ventilation as evidenced by 5 consecutive square wave end tidal carbon dioxide waveforms.

CONTACTS AND LOCATIONS:
Locations (1):
- St Johns Hospital, Livingston, United Kingdom

IPD SHARING:
Plan to Share IPD: No